CLINICAL TRIAL: NCT06558071
Title: Supplementation of Galatonol 300 mg / Striatin 30 mg Combined Bioactive Fraction in Postpartum Lactating Mothers
Brief Title: Supplementation of Galatonol 300 mg / Striatin 30 mg in Postpartum Lactating Mothers
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ASM-0120
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Lactation Induced
Keywords: Lactating mothers; Galactagogues; Galatonol /Striatin Bioactive Fraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational Group (Experimental): 1 film-coated caplet (Galatonol 300 mg/Striatin 30 mg), twice daily, after morning and evening meals
  Interventions: Drug: Galatonol 300 mg/Striatin 30 mg
- Control Group (Placebo Comparator): 1 film-coated caplet of Placebo, twice daily, after morning and evening meals
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Galatonol 300 mg/Striatin 30 mg — 1 film-coated caplet of Herba Asimor, twice daily
  Other Names: Herba Asimor
  Arms: Investigational Group
Drug: Placebo — 1 film-coated caplet of placebo Herba Asimor, twice daily
  Arms: Control Group

SUMMARY:
This is a randomized, double-blind, and placebo-controlled study involving mothers as the participant and participant's babies evaluating the effect of a 15-day-supplementation with a product containing extracts derived from a combination of herbal plants (katuk & torbangun leaves) and snakehead fish in stimulating breast milk production.

DETAILED DESCRIPTION:
The study product is a herbal product containing 300 mg Galatonol bioactive fraction, enriched with 30 mg Striatin bioactive fraction. This lactation supplement has been granted the marketing authorization from Badan Pengawas Obat dan Makanan Republik Indonesia (BPOM RI) as traditional medicine with the indication to enhance breast milk production.

A total of 160 subjects (80 subjects in each group) who have just partus, are planned to participate in this study. Eligible subjects will be allocated in a random and blinded fashion to receive one of the two products (study product or placebo) and to come for follow-up visits at Day 4, 8 and 15 (End of Study).

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to participation in the study.
2. Generally healthy women aged >= 18-35 years.
3. Having a full-term gestational age (37- 40 weeks, inclusive).
4. The infant to breastfed: having normal birth body weight (2500-4000 gr).
5. Giving consent and commitment to pursue an exclusive breastfeeding
6. Willing to comply with the study protocol.
7. Spontaneous delivery.
8. Healthy newborn baby

Exclusion Criteria:

1. Difficult breastfeeding due to organic defect;
2. Suspected COVID-19 by clinical symptoms.
3. LATCH Score < 4;
4. Choosing not to breastfeed due to other subjective or objective reasons;
5. Having multiple birth;
6. Known major medical complications during delivery;
7. Known to have breast diseases, such as: mastitis, or malignancies
8. Breastfeeding prohibited due to clindamycin injection within the past week.
9. History of smoking, alcohol drinking, or any drug abuse
10. Known to have any relevant chronic infections or illness and gestational diabetes;
11. Known to have disorders of major organs ;
12. Taking any medication or supplementation known to have galactagogue properties within the last trimester of pregnancy;
13. Taking any non-pharmacological complementary treatment within the last trimester of pregnancy aiming to affect breast milk production.
14. Participation in any other interventional clinical studies within 30 days prior to Screening.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Infant weight | Day 15
  The sufficient breastmilk supply indicated by infant weight at Day 15 of treatment (i.e. 14 days after study treatment initation) relative to Baseline (infant weight at 24 Hour post-partum).

SECONDARY OUTCOMES:
Infant weight | Day 8
  Infant weight at Day 8 of treatment (i.e. 7 days after study treatment initation) relative to Baseline.
Breastmilk production | Day 8, Day 15
  Breastmilk production at Day 8 and Day 15 of treatment (i.e. 7, and 14 days after study treatment initiation) as represented by three-hourly breast milk volume.
Breastfeeding frequency | Day 8, Day 15
  Mean breastfeeding frequency per 24 hours up to Day 8 and Day 15 of treatment (i.e. 7 and 14 days after study treatment initiation, respectively)
Prolactin level | Day 8, Day 15
  Maternal prolactin level at Day 8 and 15 of treatment
Oxytocin level | Day 8, Day 15
  Maternal oxytocin level at Day 8 and 15 of treatment
Frequency of infant void and stool | Day 8, Day 15
  Mean daily frequency of infant void and stool up to Day 8 and 15 of treatment

OTHER OUTCOMES:
Infant's daily duration of sleeping | Day 8, Day 15
  Infant's daily duration of sleeping will be evaluated as exploratory endpoint at Day 8 and 15 of treatment.
Qualitative self-assessment of breast-milk thicknes | Day 8, Day 15
  Qualitative self-assessment of breast-milk thickness will be evaluated as exploratory endpoint at Day 8 and 15 of treatment.
Body temperature | Day 8, Day 15
  Body temperature measurement as a vital sign safety parameter.
Blood pressure | Day 8, Day 15
  Blood pressure will be measured as a vital sign safety parameter.
Heart rate and respiratory rate | Day 8, Day 15
  Heart rate and respiratory rate will be measured as a vital sign safety parameter.
Random plasma glucose | Day 8, Day 15
  Random plasma glucose will be measured as a safety parameter.
Liver function | Day 15
  Liver function measurements include: serum alanine aminotransferase [ALT] and serum aspartate aminotransferase [AST].
Renal function | Day 15
  Renal function measurements include: serum creatinine
Complete blood count | Day 15
  Complete blood count measurements include: hemoglobin, hematocrit, red blood cell [RBC], white blood cell [WBC], differentiation of WBC, erythrocyte sedimentation rate [ESR], platelet count
Adverse events | Day 3, Day 8, Day 15
  Tolerability to the study product will be assessed through the evaluation of adverse events along the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Fenny Yunita, MD, MSi, PhD, Principal Investigator — Faculty of Medicine, Universitas Tarumanagara
Locations (10):
- Indonesia (10):
  - Klinik Pratama Anugrah Sleman, Sleman, Special Region of Yogyakarta
  - Private Midwife Practice (Bidan Anisa), Sleman, Special Region of Yogyakarta
  - Private Midwife Practice (Bidan Catur), Sleman, Special Region of Yogyakarta
  - Private Midwife Practice (Bidan Istri Utami), Sleman, Special Region of Yogyakarta
  - Private Midwife Practice (Bidan Istri Yuliani), Sleman, Special Region of Yogyakarta
  - Private Midwife Practice (Bidan Kisti), Sleman, Special Region of Yogyakarta
  - Private Midwife Practice (Bidan Mei), Sleman, Special Region of Yogyakarta
  - Private Midwife Practice (Bidan Tutik), Sleman, Special Region of Yogyakarta
  - Private Midwife Practice (Bidan Wati), Sleman, Special Region of Yogyakarta
  - Private Midwife Practice (Bidan Widya), Sleman, Special Region of Yogyakarta